CLINICAL TRIAL: NCT03198455
Title: Does Medicinal Mushroom Agaricus Blazei Protect Against Allergy and Asthma?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); ImmunoPharma AS (Industry)
Responsible Party: Principal Investigator, Lise Sofie Haug Nissen-Meyer, Project leader, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015/716
Record Dates: First submitted 2017-03-15; First posted 2017-06-26 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Pollen; Allergy, Asthma
MeSH Terms: conditions — Hypersensitivity; Asthma | interventions — AndoSan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Andosan (Experimental): The Agaricus blazei Murill-based mushroom extract, Andosan™, is given as one dosage 60 ml/day orally for 2 months. The intervention solution is given for 1 month's consumption at a time in a neutral plastic container
  Interventions: Dietary Supplement: Agaricus blazei Murill-based mushroom extract, Andosan™
- Placebo (Placebo Comparator): The placebo is drinking water with brownish food coloring, given as one dosage 60 ml/day orally for 2 months. The placebo solution is given for 1 month's consumption at a time in a neutral plastic container (same as for intervention/experimental solution).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Agaricus blazei Murill-based mushroom extract, Andosan™ — Dietary Supplement: Agaricus blazei Murill-based mushroom extract, Andosan™
  Arms: Andosan
Other: Placebo — Drinking water with food coloring and salt
  Arms: Placebo

SUMMARY:
Asthma and allergy is increasing in Norway and Western countries. Treatment is still mostly symptomatic. Extracts of the immunomodulatory and edible mushroom Agaricus blazei, such as Andosan™, have been shown to protect against asthma and allergy in murine models by changing the T helper cell 1(upregulation)-T helper cell 2 (downregulation) balance in the immune system. Andosan™ is produced in Japan and approved as food (mushroom juice) in Norway. Blood donors and possibly patients with pollen-derived allergy and asthma will be included in the study.The aim is to examine whether Andosan™ i) has similar clinical effects against allergy and asthma in man as it has in mice, and ii) reduces drug use and increases frequency of blood donations. Blood donors or patients who are recruited with informed consent will be given Andosan™ or placebo orally as add-on treatment to ordinary treatment for 7 weeks during the Birch pollen season, and specific IgE will be measured before, during and after the intervention, in addition to basophil activation testing and filling out of a questionnaire.

DETAILED DESCRIPTION:
Blood donors at Oslo University Hospital (OUH) Blood Bank with self-reported birch pollen allergy and/or asthma were recruited for the study during last 4 months of 2015 and first 2 months of 2016. They signed an informed consent form for the study and were randomized into Andosan™ and placebo Groups. The PI (MD) had the study key and the participants in the study were handled by other staff (nurses and bioengineers) at the blood bank. The participants were given a questionnaire that was filled out before and after the study. Before, during and after the study also blood samples were taken for allergy testing (IgE, BAT) or cytokine profiles. When the participants visited the blood bank after 3.5 weeks, they brought the study medicine vessel (plastic container) that was controlled for remaining study medicine (all should have been used) and given new study medicine for the remaining study period (3.5 weeks). The participants were also asked about possible side effects of the study medicine. In the intervention arm, Agaricus blazei-based mushroom extract Andosan™, was given, which is produced as Health food in Japan and imported as food to Norway and provided for the study by Immunopharma company, Norway. Data were collected and analyzed together after the study. Statistical help was solicited from an OUH statistician.

ELIGIBILITY:
Inclusion Criteria:

* Blood donors with birch pollen-derived allergy and asthma

Exclusion Criteria:

* Blood donors with other types of allergy and blood donors with Birch pollen allergy who are would not be in Southern Norway during most of the pollen season

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Questionnaire | Change from baseline at mid-season at approximately 3 months and after end of season at approx 6 months
  Questionnaire about allergy and asthma symptoms and medication

SECONDARY OUTCOMES:
Total IgE in serum | Change from baseline at approximately 3 months and 6 months
  Total IgE (kU/l) for all allergies
IgE anti-rBet v 1 in serum against birch pollen allergy | Change from baseline at approximately 3 months and 6 months
  Specific IgE (kUA/l) to rBet v 1 allergen
IgE anti-t3 in serum against birch pollen allergy | Change from baseline at approximately 3 months and 6 months
  Specific IgE (kUA/l) to t3 Birch pollen extract
Basophil Activation Test (BAT) | Change from baseline at approximately 3 months and 6 months
  Basophil granulocytes are isolated from venous blood samples of study participants
Cytokines in serum | Change from baseline at approximately 6 months
  Th1, Th2, pro-and anti-inflammatory cytokines (pg/ml) in plasma was measured by Luminex multi cytokine kit analysis

IPD SHARING:
Plan to Share IPD: Undecided